CLINICAL TRIAL: NCT01696760
Title: Aspirin and Compression Devices for VTE Prophylaxis in Orthopaedic Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Joel Mayerson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-10055; NCI-2012-00894 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Bone Metastases; Musculoskeletal Cancer; Soft Tissue Sarcoma; Thromboembolism
MeSH Terms: conditions — Sarcoma; Thromboembolism | interventions — Aspirin; Enoxaparin; enoxaparin sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (acetylsalicylic acid and PCD) (Experimental): Patients receive acetylsalicylic acid orally PO BID and wear PCD on days 1-28 after surgery.
  Interventions: Drug: acetylsalicylic acid; Device: PCD
- Arm II (enoxaparin and PCD) (Experimental): Patients receive enoxaparin subcutaneously SC QD and wear PCD on days 1-28 after surgery.
  Interventions: Drug: enoxaparin; Device: PCD

INTERVENTIONS:
Drug: acetylsalicylic acid — 325 mg twice a day
  Other Names: ASA; Ecotrin; Empirin; Extren
  Arms: Arm I (acetylsalicylic acid and PCD)
Drug: enoxaparin — 40 mg once daily
  Other Names: Enoxaparin Sodium; Lovenox
  Arms: Arm II (enoxaparin and PCD)
Device: PCD — Wear PCD (Flowtron calf compression). Patients will continue to use PCDs for the duration of their hospitalization. If patients refuse to wear the PCDs, they will be withdrawn from the study.
  Other Names: thromboembolism prophylaxis; Flowtron calf compression

SUMMARY:
This is a research study to compare the efficacy of aspirin (acetylsalicylic acid) and pneumatic compression devices versus enoxaparin (also known as Lovenox) and pneumatic compression devices in preventing deep vein thrombosis in patients with pelvic and lower extremity malignant tumors and undergoing surgery. Pneumatic compression devices are also known as sequential compression devices and are inflatable compression sleeves that are placed around patient's legs to reduce the risk of clot formation deep vein thrombosis. Pneumatic compression devices are made of a soft material that wraps around the lower leg and periodically squeeze the calf. A deep vein thrombosis is a blood clot. Most hospitalized patients wear these as a preventive measure. Pneumatic compression devices alone are not sufficient to prevent deep vein thrombosis formation. Therefore, medicines, such as aspirin and enoxaparin are utilized. Both drugs are used for prevention, but there are no studies in patients with musculoskeletal tumors which have determined whether one drug is better than another. The knowledge gained from this study will determine whether aspirin and pneumatic compression devices is the same or better than enoxaparin and pneumatic compression devices in preventing deep vein thrombosis in this patient population and may result in fewer wound and bleeding complications

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform a randomized prospective study to determine efficacy of acetylsalicylic acid (ASA)+pneumatic compression device (PCD) prophylaxis compared to low-molecular weight heparin (LMWH)+PCD in patients undergoing orthopaedic procedures for musculoskeletal neoplasms (MSN) of the pelvis and lower extremity.

II. To prove that ASA+PCD is clinically equivalent to or better than LMWH+PCD in providing deep vein thrombosis (DVT) prophylaxis in this patient population and results in fewer major bleeding complications.

III. To measure rates of postoperative DVT and pulmonary embolism (PE) as primary outcomes.

SECONDARY OBJECTIVES:

I. To measure secondary outcomes including rates of readmission, reoperation, bleeding complications (including hematoma formation and prolonged wound drainage), and death.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive acetylsalicylic acid orally (PO) twice daily (BID) and wear PCD on days 1-28 after surgery.

ARM II: Patients receive enoxaparin subcutaneously (SC) once daily (QD) and wear PCD on days 1-28 after surgery.

After completion of study treatment, patients are followed up at 2 weeks, 6 weeks, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

-Scheduled or to be scheduled for surgery performed on neoplasms of the pelvis or lower limbs, including both primary musculoskeletal lesions as well as metastatic lesions; these neoplasms may include major tumor resections, metastatic and pathologic fractures of the hip and lower extremities (LE), open biopsies, and primary malignant tumors; an active malignant neoplasm must be present at the time of surgery

Exclusion Criteria:

* Prior history of DVT or PE
* Previously placed vena cava filter
* No detectable malignant disease at the time of operation
* Previous arterial thrombosis (myocardial infarction [MI], cerebral vascular accident [CVA])
* Severe platelet dysfunction (uremia, medications, dysplastic hematopoiesis); excluded if platelets < 50,000
* Preoperative anticoagulation or active/serious bleeding in past 2 weeks (prothrombin time [PT] & partial thromboplastin time [PTT] > 1.6 & > 35)
* Hypersensitivity or allergy to aspirin or heparin (including those diagnosed with heparin-induced thrombocytopenia)
* Conditions associated with bleeding (active ulcer disease, recent neurosurgery, bleeding disorders)
* Patients with renal insufficiency (creatinine [Cr] > 1.5)
* Pregnant patients
* Epidural anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Mayerson, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Started | 9 | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD) | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 11
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: DVT Incident Rate
Description: This study will test if the ASA+PCD treatment group has a DVT rate (P1) not more than the DVT rate of the LMWH+PCD treatment group (P0) using a one sided test for these two proportions. Statistical significance will be defined as p < 0.05.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

2. Secondary Outcome: Pulmonary Embolism Rate
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

3. Secondary Outcome: Development of Other Complications (Including Bleeding Complications)
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

4. Secondary Outcome: Readmission Rate to Hopsital
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

5. Secondary Outcome: Hematoma Formation
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

6. Secondary Outcome: Excessive Wound Drainage
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

7. Secondary Outcome: Death Rate
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Acetylsalicylic Acid and PCD) | Arm II (Enoxaparin and PCD)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/9 | 0/3

LIMITATIONS AND CAVEATS:
Overall patient compliance for the study was low

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes